CLINICAL TRIAL: NCT00262249
Title: Effect of Growth Hormone in Children With Growth Hormone Deficiency and Idiopathic Short Stature
Brief Title: Effect of Growth Hormone in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGH-2051
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Growth Disorder; Idiopathic Short Stature
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of the trial is to compare the effect of Norditropin® using different dosing regimens in children suspected of growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected GHD
* Height < -2.0 SDS
* Serum IGF-I less than or equal to -1.0 SDS
* Bone age less than or equal to 9 years for boys and less than or equal to 7 years for girls.
* Puberty Tanner Stage I

Exclusion Criteria:

* Previous use of growth hormone
* Growth retardation attributable to causes other than GHD (e.g. inborn errors of metabolism, primary bone disease, chromosomal disorders, etc.)
* Intrauterine growth retardation: birth weight < 3rd percentile.
* Administration of other growth-altering medications.
* Evidence of any malignancy or intracranial tumors.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2000-08; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change in height standard deviation score | 24 month

SECONDARY OUTCOMES:
IGF-I
IGFBP-3
free IGF-I

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (37):
- United States (37):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Stanford, California
  - Novo Nordisk Investigational Site, New Haven, Connecticut
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Morristown, New Jersey
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Stony Brook, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Cohen P, Rogol AD, Howard CP, Bright GM, Kappelgaard AM, Rosenfeld RG; American Norditropin Study Group. Insulin growth factor-based dosing of growth hormone therapy in children: a randomized, controlled study. J Clin Endocrinol Metab. 2007 Jul;92(7):2480-6. doi: 10.1210/jc.2007-0204. Epub 2007 Mar 13. PMID 17356043
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com